CLINICAL TRIAL: NCT02077400
Title: The Use of Prophylactic Antibiotic in Treatment of Fingertip Amputation: A Randomized Prospective Trial
Brief Title: Prophylactic Antibiotic in Treatment of Fingertip Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, guy rubin, Dr., HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0115-09-EMC
Record Dates: First submitted 2014-03-02; First posted 2014-03-04 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Infection Rate After Fingertip Amputation
MeSH Terms: interventions — Cefazolin

ARMS (2):
- no antibiotic (No Intervention)
- Cephazolin (Active Comparator): cefazoline
  Interventions: Drug: Cephazolin

INTERVENTIONS:
Drug: Cephazolin — Cephazolin
  Other Names: Cefamezine
  Arms: Cephazolin

SUMMARY:
Fingertip amputation is a common injury. Considerable controversy exists as to whether prophylactic antibiotics are necessary for this injury. The investigators goal was to compare the rate of infections among subgroups with and without prophylactic antibiotic treatment. The study hypothesis was that infection rates were similar in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* fingertip amputation with bone exposed

Exclusion Criteria:

* under the age of 18 years
* if the patient had diabetes
* oncological disorder
* immune deficiency
* bleeding disorder
* used steroids regularly
* presented with a grossly contaminated wound or other injury requiring antibiotic treatment
* were currently taking antibiotics, or had a previous allergic reaction to cephalosporins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
infection rate | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek medical center, Afula, Israel